CLINICAL TRIAL: NCT01207167
Title: Mediators of Atherosclerosis in South Asians Living in America
Acronym: MASALA
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Northwestern University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); New York University (Other)
Responsible Party: Sponsor
Other Study IDs: MASALA; R01HL093009 (NIH); R01MD016071 (NIH); R01HL149809 (NIH)
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Coronary Artery Disease; Coronary Disease
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
South Asian (Indian, Pakistani, Bangladeshi, Nepali, and Sri Lankan) individuals have high rates of cardiovascular disease that is not explained by traditional cardiovascular risk factors. Though South Asians represent over one-quarter of the world's population, there are no longitudinal studies in this high-risk ethnic group. The investigators aim to establish a longitudinal study of South Asians at three United States centers to identify risk factors linked to subclinical atherosclerosis and incident cardiovascular disease. The purpose of this study is to understand the causes of heart disease and stroke in South Asians and compare these causes to those in other United States ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* South Asian ancestry defined by having at least 3 grandparents born in one of the following countries: India, Pakistan, Bangladesh, Nepal, or Sri Lanka
* age between 40 and 84 years.

Exclusion Criteria:

* Physician diagnosed heart attack, stroke or transient ischemic attack (TIA), heart failure, or angina (or use of nitroglycerin)
* Current atrial fibrillation
* Past history of cardiovascular procedures (coronary artery bypass graft (CABG) Surgery, angioplasty, valve replacement, pacemaker or defibrillator implantation, or any surgery on the heart or arteries)
* Active treatment for cancer
* Life expectancy less than 5 years due to serious medical illness
* Impaired cognitive ability as judged by the reviewer
* Plans to move out of the study region in next 5 years
* Weight greater than 300 pounds
* Living in a nursing home or on a waiting list
* Unable to speak/read/write English, Hindi, Urdu, or Bangla

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: South Asians (individuals from India, Pakistan, Nepal, Bangladesh, and Sri Lanka) adults between the ages of 40 and 84 years without cardiovascular disease living in the San Francisco Bay Area, Chicago Area, or New York City Area.
Sampling Method: Probability Sample
Enrollment: 2314 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Coronary artery calcium prevalence in South Asians | Baseline

SECONDARY OUTCOMES:
Carotid intima media thickness | Baseline
Diabetes Prevalence | Baseline
Change from baseline Coronary artery calcium prevalence in South Asians at 4 years | Baseline to Year 4
Incidence of type 2 diabetes after approximately 4 years of follow-up | Baseline to Year 4

CONTACTS AND LOCATIONS:
Overall Officials: Alka Kanaya, MD, Principal Investigator — University of California, San Francisco; Namratha Kandula, MD, Principal Investigator — Northwestern University; Nadia Islam, PhD, Principal Investigator — New York University
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - New York University, New York, New York

IPD SHARING:
Plan to Share IPD: No